CLINICAL TRIAL: NCT04615026
Title: Prevalence of Thrombosis in COVID-Patients in Correlation to Humoral and Cellular Immunity
Brief Title: Prevalence of Thrombosis in COVID-Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Responsible Party: Principal Investigator, Alexander Hyhlik-Dürr, Head of department, University Hospital Augsburg
Other Study IDs: COVID Thrombose
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Aliquots for proteomics analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID 19 patients: all patients with positive SARS-CoV 2 swap
  Interventions: Diagnostic Test: duplex sonography

INTERVENTIONS:
Diagnostic Test: duplex sonography — all patients with consent receive a duplex ultrasound, blood test, cognitive test and test of smelling
  Other Names: test of smell; cognitive test; blood sample

SUMMARY:
Examination of the prevalence of thrombosis in COVID-patients, especially in an out-patient setting. Assessment by duplex sonography. If thrombosis is detected, we will correlate it with immunity status. Assessment of health issues and cognitive function as late complication after infection.

ELIGIBILITY:
Inclusion Criteria:

* SARS CoV 2 positive swap, at least 4 weeks after infection

Exclusion Criteria:

* under 18 years old no consent anemia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all SARS CoV 2 positive patients registered at local health departments (Augsburg) are invited to join the study
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
prevalence of thrombosis | 20 minutes

SECONDARY OUTCOMES:
correlation to immunity | 20 minutes
Assessment of late complications | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hyhlik-Duerr, MD, Principal Investigator — University Hospital Augsburg
Locations (1):
- University Hospital Augsburg, Augsburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
data as pseudonyms

REFERENCES:
- [Derived] Schmidbauer L, Kirchberger I, Gosslau Y, Warm TD, Hyhlik-Durr A, Linseisen J, Meisinger C. The association between the number of symptoms and the severity of Post-COVID-Fatigue after SARS-CoV-2 infection treated in an outpatient setting. J Neurol. 2023 Jul;270(7):3294-3302. doi: 10.1007/s00415-023-11752-9. Epub 2023 May 23. PMID 37219607